CLINICAL TRIAL: NCT01250977
Title: The Effect of Acetylcholinesterase Inhibitors on Smoking Behavior
Brief Title: Effect of Donepezil on Smoking
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: UPCC 12910
Record Dates: First submitted 2010-10-20; First posted 2010-12-01 (Estimated); Results first posted 2019-07-11 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Smoking
Keywords: Non-treatment seeking smokers, reporting consumption of at least; 10 cigarettes per day for at least the past 6 months
MeSH Terms: conditions — Smoking | interventions — Donepezil

STUDY DESIGN:
Intervention Model Description: This is a double-blind, human laboratory study using a between-subject design between smokers who are randomized to either donepezil HCL (Aricept®) (n=15) or placebo (n=15) for 4 weeks. Treatment randomization will be done to match both groups for age and sex.
Who Masked: Participant, Investigator
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Participants are instructed to take one placebo pill every night before going to bed with a glass of water for 28 days.
  Interventions: Drug: Placebo
- Donepezil (Experimental): Participants are instructed to take one 5mg pill (donepezil HCL [Aricept®]) every night before going to bed with a glass of water for 28 days.
  Interventions: Drug: Donepezil

INTERVENTIONS:
Drug: Donepezil
  Other Names: Aricept
  Arms: Donepezil
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objective of this proof-of-concept pilot study is to evaluate Donepezil HCL (Aricept) for side effects and effects on smoking behavior and performance on neurocognitive tasks in a population of dependent smokers.

DETAILED DESCRIPTION:
Nicotine dependence is a major public health problem and currently available treatments are ineffective for the majority of smokers. Thus, there is a need to develop and test novel medications to assist smokers to quit smoking. This pilot feasibility study examined: (1) tolerability and medication adherence, and (2) the effects of donepezil versus placebo on smoking behavior and cognitive performance in non-treatment seeking smokers. We predicted that 4 weeks of donepezil would improve working memory at the highest task difficulty level and sustained attention. Because participants in this study were not trying to quit, change in smoking behavior was a secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

* 30 smokers ages 18-50 who have smoked at least 10 cigarettes per day for the past 6 months, will be eligible to participate. They must be able to provide informed consent.

Exclusion Criteria:

* Smoking Behavior:

  1. Current enrollment or plans to enroll in a smoking cessation program, or use other smoking cessation medications in the next 2 months.
  2. Provide a CO reading less than 10 ppm at medical screening.
  3. Participants who roll their own cigarettes.
  4. Regular use of chewing tobacco or snus.
* Alcohol/Drugs 1) History of substance abuse and/or currently receiving treatment for substance abuse (e.g. alcohol, opioids, cocaine, marijuana, or stimulants). 2) Current alcohol consumption that exceeds 25 standard drinks/week. 3) Providing a breath alcohol concentration (BrAC) reading of greater than or equal to 0.01 at medical screen, baseline, or testing sessions.
* Medical:

  1. Women who are pregnant, planning a pregnancy, or lactating; all female subjects shall undergo a urine pregnancy test prior to enrollment and must agree in writing to use an approved method of contraception.
  2. Lifetime history or current diagnosis of psychosis, bipolar disorder, anxiety disorder, or schizophrenia, as identified by the MINI. Individuals with a past history of depression are eligible as long as their major depression episode was more than 6 months ago.
  3. Serious or unstable disease within the past 6 months i.e. heart disease, liver/kidney failure)
  4. Other medical conditions such as peptic ulcer disease; beign prostatic hypertrophy or bladder outflow problems; asthma or chronic obstructive pulmonary disease.
  5. BP reading of 170/100 at medical screening session.
* Medication:

  1) Current use, recent discontinuation within last 14 days or planned use of the following medications:
* Any form of smoking cessation medication, i.e. Zyban, Wellbutrin, Wellbutrin SR, Chantix, nicotine replacement therapy
* Psychotropic medications (anti-psychotics, anti-depressants, anti-anxiety or anti-panic medications, mood stabilizers and stimulants)
* Current treatment with other acetylcholinesterase inhibitors (ACIs) like donepezil HCL (Aricept), tacrine, rivgastigmine and galantamine
* Anti-seizure meds, and other meds that affect the cholinergic system such as mecamylamine, atropine, succinylcholine, ketocaonazole, quinidine, bethanechol, iprapropium, bromide, dicyclomine, benztropine, carisprodol, zantac, and procardia.

  2) Patients shallbe instructed to refrain from using any study prohibited drugs (note participants are allowed to take prescription medicines not in the exclusion list)throughout their participation in the study.
* Other

  1. Inability to complete the baseline study procedures within thee hours and/or correctly, as determined by the PI.
  2. Non-English speakers.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-01-11 (Actual); Primary Completion 2011-12-06 (Actual); Study Completion 2011-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Strasser, MBBS, PhD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty subjects were consented and screened for eligibility at an Intake Visit at the Center for Interdisciplinary Research on Nicotine Addiction (Philadelphia, PA).
Pre-assignment Details: Twenty subjects ultimately completed a Baseline Visit and were randomized to receive Donepezil or Placebo.
Period: Overall Study
Arm/Group | Placebo | Donepezil
Started | 6 | 14
Completed | 6 | 12
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Population: All participants receiving at least one dose of Donepezil or Placebo are included in the analysis population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Donepezil | Total
Number analyzed (Participants) | 6 | 14 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 14 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.00 (9.58) | 33.24 (10.51) | 33.75 (9.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 4 | 9 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 14 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 5 | 5
  White | 5 | 8 | 13
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 14 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in True Positives on the 3-Back Level of the Letter-N-Back Neurocognitive Task at Day 28 (i.e., Week 4)
Description: Neurocognitive task performance was assessed during baseline and each testing day (Day 7, 14, 21, and 28) using computerized tasks. Working memory was assessed with the Letter-N-back task.
Time Frame: Baseline and Day 28
Measure: Mean (Standard Error); unit: True positive responses
Arm/Group | Placebo | Donepezil
Number analyzed (Participants) | 6 | 12
True positive responses | .59 (.88) | 3.4 (.88)

2. Primary Outcome: Change From Baseline in Discriminability on the Penn Continuous Performance Neurocognitive Task at Day 28 (i.e., Week 4)
Description: Sustained attention was assessed with the Penn Continuous Performance Task (P-CPT). The primary outcome measure was the change from Baseline in discriminability (score) on the P-CPT at Day 28. The discriminability score is the mathematical difference between the total correct (i.e., true positives and correct non-responses) and incorrect (i.e., errors of commission and omission) responses to a series of stimuli presented during the P-CPT. The unit of measure is number of correct responses less the number of incorrect responses. A higher discriminability score at a single time point indicates a better performance on the P-CPT. A positive change in discriminability score between Baseline and Day 28 indicates improved performance over time. In its purest mathematical sense, the discriminability measure is a difference of difference scores and therefore is without scale limits, that is, there are no minimum or maximum values one could theoretically obtain.
Time Frame: Baseline and Day 28
Measure: Mean (Standard Error); unit: correct minus incorrect responses
Arm/Group | Placebo | Donepezil
Number analyzed (Participants) | 6 | 12
correct minus incorrect responses | -.1 (.08) | .5 (.08)

3. Secondary Outcome: Change From Baseline in Smoking Behavior (i.e., Cigarettes Per Day) at Day 28 (i.e., Week 4)
Description: At each visit, smoking rate (i.e., cigarettes per day) was assessed using standard Timeline Followback methods. Weekly averages were computed to assess group differences in changes in smoking behavior from Baseline to Day 28.
Time Frame: Baseline and Day 28
Measure: Mean (Standard Error); unit: cigarettes per day
Arm/Group | Placebo | Donepezil
Number analyzed (Participants) | 6 | 12
cigarettes per day | 3.3 (4.4) | 1.9 (1.0)

4. Secondary Outcome: Summary Side Effect Score at Day 28 (i.e., Week 4)
Description: A 38-item self-report measure of the side effects associated with Donepezil (e.g., nausea) was administered to all participants at observation and testing days through Day 28. For each item, side effect severity was rated on a 4-point scale (0 = not present, 1 = mild, 2 = moderate, 3 = severe). The side effect summary score from the measure collected at Day 28 was considered the dependent measure because Day 28 is when the medication reached steady state. The side effect summary score was calculated by taking the mean score (i.e., sum of all 38 items [each item rated on a scale 0-3] divided by 38) of the measure from each participant at Day 28, adding the means, and then dividing the sum of the means by the number of participants within each group. A higher summary score indicates a higher general incidence rate and severity of side effects.
Time Frame: Day 28
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Donepezil
Number analyzed (Participants) | 6 | 12
score on a scale | 2.3 (.7) | 1.1 (.5)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over a 28-day period.
Description: The safety population described within this section includes all subjects who received at least one dose of Donepezil or Placebo.
  Systematic Assessment: Side effect severity was rated on a 4-point scale (0 = not present, 1 = mild, 2 = moderate, 3 = severe) using a 38-item self-report measure based on common side effects of Donepezil (e.g., nausea) at all in-person visits (n=9).
Arm/Group | Placebo | Donepezil
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/14
Other Adverse Events (participants affected / at risk) | 5/6 | 14/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=6) | Donepezil (N=14)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (10)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 4 (8)
Insomnia (Psychiatric disorders) | 2 (10) | 4 (10)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Muscle Cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (3)
Fatigue or tiredness (General disorders) | 4 (14) | 6 (13)
Decreased Appetite (General disorders) | 0 (0) | 6 (10)
Headache (Nervous system disorders) | 3 (16) | 5 (17)
Body Pain (including Back Pain) (Musculoskeletal and connective tissue disorders) | 1 (3) | 3 (7)
Large Bruises (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Weight Decrease (General disorders) | 0 (0) | 3 (6)
Joint Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (14)
Dizziness (General disorders) | 2 (4) | 3 (7)
Depressed Mood (Psychiatric disorders) | 1 (1) | 1 (4)
Abnormal Dreams (Psychiatric disorders) | 3 (9) | 8 (21)
Frequent Urination (Renal and urinary disorders) | 0 (0) | 4 (7)
Drowsiness (General disorders) | 3 (15) | 7 (11)
Chest Pain (Cardiac disorders) | 1 (1) | 2 (3)
Hostility (Psychiatric disorders) | 0 (0) | 1 (3)
Nervousness (Psychiatric disorders) | 1 (6) | 1 (4)
Confusion (Psychiatric disorders) | 1 (1) | 2 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (12) | 6 (18)
Itching (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (5)
Abnormal Vision (Eye disorders) | 0 (0) | 1 (3)
Eye Redness/Irritation (Eye disorders) | 1 (1) | 4 (10)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 5 (14)
Dehydration (General disorders) | 2 (8) | 3 (6)
Incontinence (Renal and urinary disorders) | 0 (0) | 1 (4)
Abdominal pain or bloating (Gastrointestinal disorders) | 1 (1) | 2 (3)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (3)
Fever (General disorders) | 0 (0) | 2 (3)
Hot Flashes (General disorders) | 0 (0) | 1 (4)
Black Stool (Gastrointestinal disorders) | 0 (0) | 1 (1)
Difficulty Urinating (Renal and urinary disorders) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes